CLINICAL TRIAL: NCT06121791
Title: Establishment Reference Values for Abdominal Skeletal Muscle Compartments in Turkish Children
Brief Title: Abdominal Skeletal Muscle Compartments in Turkish Children
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Aydın, Researcher, Assoc Prof, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPMR-ct-mscl-chld
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Child Development; Sarcopenia
Keywords: children; Abdominal Skeletal Muscle; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Normal values of abdominal level muscle areas of Turkish children — age, sex, L3-L4 LEVEL: Psoas muscle area, Paraspinal muscle area, Abdominal muscle area, L4-L5 LEVEL: Psoas muscle area, Paraspinal muscle area, Abdominal muscle area

SUMMARY:
The aim of this study was to establish reference values for three compartments of the abdominal skeletal muscle area (psoas muscle area, paraspinal muscle area, and total skeletal muscle area) obtained from cross-sectional Computed tomography images in Turkish Children

DETAILED DESCRIPTION:
The aim in this study is to determine reference values for Turkish children by evaluating the abdominal region skeletal muscle area (psoas muscle, paraspinal muscles and total skeletal muscle in the section) obtained from cross-sectional CT images.

Material Method of the Research The study was planned as a retrospective study. Patients under 18 years of age who are admitted to Istanbul Province Bağcılar Training and Research Hospital with acute abdominal pain or acute trauma between May 5, 2017 and May 5, 2023 and who underwent abdominal computed tomography (CT) imaging on this date of application will be scanned through the hospital information management system. Past diagnoses of these patients will be questioned and those with chronic diseases will be excluded from the study.

CT images of the patients will be retrieved from the PACS database. From the sections taken at the L3-L4, L4-L5 levels, the cross-sectional area of the psoas muscle, paraspinal muscles and the total skeletal muscles in that section will be measured using the hospital's SYNAPS system. The results will be recorded in cm2.

ELIGIBILITY:
Inclusion Criteria:

* No chronic disease
* Being under 18 years of age
* Being Turkish
* Determining that an abdominal CT was performed in the hospital records

Exclusion Criteria:

* Patients with malignancy or known chronic disease
* Patients with mental health problems

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Healthy Turkish children
Sampling Method: Non-Probability Sample
Enrollment: 2168 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
L3-L4 LEVEL: Psoas muscle area | 1 interview day
  The Psoas muscle area at the L3-L4 vertebra level in the patients' abdominal computed tomography will be measured.
L3-L4 LEVEL:Paraspinal muscle area | 1 interview day
  The Paraspinal muscle area at the L3-L4 vertebra level in the patients' abdominal computed tomography will be measured.
L3-L4 LEVEL: Abdominal muscle area, | 1 interview day
  The Abdominal muscle area at the L3-L4 vertebra level in the patients' abdominal computed tomography will be measured.
L4-L5 LEVEL: Psoas muscle area | 1 interview day
  The Psoas muscle area at the L4-L5 vertebra level in the patients' abdominal computed tomography will be measured.
L4-L5 LEVEL: Paraspinal muscle area | 1 interview day
  The Paraspinal muscle area at the L4-L5 vertebra level in the patients' abdominal computed tomography will be measured.
L4-L5 LEVEL: Abdominal muscle area, | 1 interview day
  The Abdominal muscle area at the L3-L4 vertebra level in the patients' abdominal computed tomography will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital; EDA CINGOZ, Principal Investigator — ISTANBUL BAĞCILAR TRAINING AND RESEARCH HOSPITAL RADIOLOGY UNIT
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kudo W, Terui K, Hattori S, Takenouchi A, Komatsu S, Oita S, Sato Y, Hishiki T. Establishment and validation of reference values for abdominal skeletal muscle compartments in children. Clin Nutr. 2023 May;42(5):653-660. doi: 10.1016/j.clnu.2023.02.022. Epub 2023 Mar 2. PMID 36934494
- [Background] Harbaugh CM, Zhang P, Henderson B, Derstine BA, Holcombe SA, Wang SC, Kohoyda-Inglis C, Ehrlich PF. Personalized medicine: Enhancing our understanding of pediatric growth with analytic morphomics. J Pediatr Surg. 2017 May;52(5):837-842. doi: 10.1016/j.jpedsurg.2017.01.030. Epub 2017 Jan 29. PMID 28189451
- [Background] Metzger GA, Sebastiao YV, Carsel AC, Nishimura L, Fisher JG, Deans KJ, Minneci PC. Establishing Reference Values for Lean Muscle Mass in the Pediatric Patient. J Pediatr Gastroenterol Nutr. 2021 Feb 1;72(2):316-323. doi: 10.1097/MPG.0000000000002958. PMID 33003166
- [Background] Lurz E, Patel H, Lebovic G, Quammie C, Woolfson JP, Perez M, Ricciuto A, Wales PW, Kamath BM, Chavhan GB, Juni P, Ng VL. Paediatric reference values for total psoas muscle area. J Cachexia Sarcopenia Muscle. 2020 Apr;11(2):405-414. doi: 10.1002/jcsm.12514. Epub 2020 Jan 9. PMID 31920002